CLINICAL TRIAL: NCT06146855
Title: Amnion Membrane as a Soft Tissue Substitute Versus De- Epithelialized Free Gingival Graft Using the Tunneling Technique in Management of Gingival Recession Defects: A Randomized Controlled Clinical Trial.
Brief Title: Amnion Membrane Versus DFGG Using the Tunneling Technique in Management of Gingival Recession Defects.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mashaly, Assistant lecturer of Periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMvsDFGG
Record Dates: First submitted 2023-11-18; First posted 2023-11-27 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tunneling with amnion membrane (Experimental)
  Interventions: Procedure: Tunneling procedure with Amnion Membrane
- Tunneling with De-epithelialized Free Gingival Graft (Active Comparator)
  Interventions: Procedure: Tunneling procedure with De-epithelialized Free Gingival Graft

INTERVENTIONS:
Procedure: Tunneling procedure with Amnion Membrane — Root Coverage by tunneling procedure with the addition of Amnion Membrane as a soft tissue substitute
  Arms: Tunneling with amnion membrane
Procedure: Tunneling procedure with De-epithelialized Free Gingival Graft — Root Coverage by tunneling procedure with the addition of De-epithelialized Free Gingival Graft
  Arms: Tunneling with De-epithelialized Free Gingival Graft

SUMMARY:
Treatment of gingival recession is indicated mainly for esthetic reasons and keratinized tissue augmentation (Zucchelli and Mounssif, 2015). An array of surgical techniques has been proposed by the literature to cover gingival recession defects with well-documented successful outcomes. The selection of one technique over the other depends on many factors. Some of these factors are related to the gingival recession defect itself, others are related to the anatomy of the palatal fibromucosa, or related to the patient variabilities (Zucchelli and De Sanctis, 2000).

Controversy exists in the literature regarding the patient morbidity after connective tissue graft harvesting. Inconclusive postulations have been made about the post-operative patient morbidity outcomes and root coverage outcomes when comparing connective tissue graft harvesting in comparison to allograft membranes used for root coverage.

The use of connective tissue graft in combination with root coverage techniques remain the gold standard for root coverage procedures. The problem with the connective tissue graft is that harvesting a graft from the palate increases morbidity, needs an extra surgical site which is more traumatic for the patient, depends on the donor tissue which could be limited, increases surgical chair-time and needs increased surgical skills (Cortellini & Pini Prato 2012).

The rationale behind the use of amnion membrane is to avoid the morbidity inherent with connective tissue graft harvesting.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* Periodontally and systemically healthy.
* Presence of RT1 or RT2 buccal gingival recession defects ≥2 mm in depth.
* Full-mouth plaque and bleeding score of <15% and no probing depths >3 mm.
* Absence of non-carious cervical lesions (NCCLs) and non-detectable cemento-enamel junction (CEJ) at the defect sites.

Exclusion Criteria:

* RT3 recession defects.
* Smokers as smoking is a contraindication for any plastic periodontal surgery (Khuller, 2009).
* Presence of caries lesions or restorations in the cervical area.
* Intake of medications which impede periodontal tissue health and healing.
* Medical contraindications for periodontal surgical procedures.
* Uncooperative patients not willing to complete the follow up period.
* Pregnancy and lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Recession depth | 3-6 month
  Measured from the CEJ to the most apical extension of the gingival margin.

SECONDARY OUTCOMES:
Recession width | 3-6 month
  Measured horizontally between the borders of the recession.
Percentage of root coverage | 6 months
  (Preoperative vertical recession - Postoperative vertical recession/preoperative vertical recession) x 100.
Root coverage esthetic score | 6 months
  Based on Cairo et al., (2009) the root coverage esthetic score (RES) system evaluated five variables 6 months following surgery: gingival margin (GM), marginal tissue contour (MTC), soft tissue texture (STT), MGJ alignment, and gingival color (GC).
Gingival Thickness | 3-6 months
  Determined 2 mm apical to the gingival margin with a short needle for anesthesia and a 3 mm diameter silicon disk stop. The needle is inserted perpendicular to the mucosal surface, through the soft tissues with light pressure until a hard surface is felt. The silicon disk stop is then placed in tight contact with the soft tissue surface with the coronal border overlapping the soft tissue margin. As the needle is located in the center of the silicon disk, measurement of GT is performed 2 mm apical from the gingival margin. After careful removal of the needle, the penetration depth is measured with a caliper accurate to the nearest 0.1 mm (Paolantonio et al., 2002; da Silva et al., 2004; Joly et al., 2007).
Keratinized tissue width | 3-6 months
  Measured as the distance between the gingival margin and the mucogingival junction (MGJ).
Post-Operative Pain | 1 week
  Visual Analogue Scale (VAS) with numbers from 0 to 10 ('no pain' to 'worst pain imaginable') measured daily for the first week postoperatively.
Post-Surgical Patient Satisfaction | 1 week
  A 3-item questionnaire is asked and the patients shall use a 7- point answer scale. (Kiyak et al., 1984)
Surgical time | intraoperative
  Total time of the surgical procedure measured using a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mashaly, MSc, Principal Investigator — Assistant lecturer of Periodontology, Cairo University; Noha Ghallab, Phd, Study Chair — Professor of Oral Medicine and Periodontology, Cairo University; Weam El Battawy, Phd, Study Director — Assistant Professor of Oral Medicine and Periodontology, Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Bakhishov H, Isler SC, Bozyel B, Yildirim B, Tekindal MA, Ozdemir B. De-epithelialized gingival graft versus subepithelial connective tissue graft in the treatment of multiple adjacent gingival recessions using the tunnel technique: 1-year results of a randomized clinical trial. J Clin Periodontol. 2021 Jul;48(7):970-983. doi: 10.1111/jcpe.13452. Epub 2021 Apr 7. PMID 33751615
- [Background] Ghahroudi AA, Khorsand A, Rokn AR, Sabounchi SS, Shayesteh YS, Soolari A. Comparison of amnion allograft with connective tissue graft for root coverage procedures: a double-blind, randomized, controlled clinical trial. J Int Acad Periodontol. 2013 Oct;15(4):101-12. PMID 24364174